CLINICAL TRIAL: NCT01040884
Title: A Prospective, Open-Label, Single-Arm, Single-Center Study Evaluating the Preliminary Safety and Accuracy of the ActiSight™ Needle Guidance System in Patients Undergoing CT-Guided Percutaneous Aspiration, Biopsy and RF Ablations
Brief Title: Safety And Accuracy Study Of The Actisight™ Needle Guidance System In Patients Undergoing CT-Guided Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ActiViews Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASNG-LFNA-101-IL-H
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ActiSight Needle Guidance System (Experimental): ActiSight™ Needle Guidance System is comprised of several sub-system components: a computer, a disposable ActiSensor optical sensor, and the disposable ActiSticker, which provides a reference for the insertion of the tool and for the camera.
  Interventions: Other: ActiSight Needle Guidance System

INTERVENTIONS:
Other: ActiSight Needle Guidance System — ActiSight™ Needle Guidance System is comprised of several sub-system components: a computer, a disposable ActiSensor optical sensor, and the disposable ActiSticker, which provides a reference for the insertion of the tool and for the camera
  Other Names: ActiSensor; ActiSticker

SUMMARY:
This will be a prospective, single-arm, single-center, open-label study to evaluate the preliminary safety and accuracy of the ActiSight™ Needle Guidance System in patients undergoing CT-guided percutaneous aspiration and RF Ablations The procedure will be performed by a trained physician. Subjects will be screened for inclusion in the study. Following signing of informed consent, screening procedures will be performed including demographic and medical history, vital signs, anthropometrics), chest radiography, if applicable and CT scanning, blood samples for coagulation indices (PT, APTT), if applicable, and pregnancy test in women of child-bearing potential.

Within an 18-day screening period, eligible subjects will be enrolled into the study and undergo percutaneous aspiration or percutaneous biopsy or RF ablation utilizing the ActiSight™ Needle Guidance system using CT to guide the needle. Subjects will be followed-up for at least one hour at the clinic for safety and preliminary accuracy evaluations. An erect chest radiograph will be performed within 90 minutes of observation after chest aspiration if performed to detect the majority of post procedure pneumothoraces for biopsies in the chest. Post procedural CT will be performed according to the physician's consideration. ** Note ** If any complications are observed while using the ActiSight System, the investigator will revert to using standard procedure.

DETAILED DESCRIPTION:
Within an 18-day screening period, eligible subjects will be enrolled into the study and undergo percutaneous aspiration or percutaneous biopsy or RF ablation utilizing the ActiSight™ Needle Guidance system using CT to guide the needle. Subjects will be followed-up for at least one hour at the clinic for safety and preliminary accuracy evaluations. An erect chest radiograph will be performed within 90 minutes of observation after chest aspiration if performed to detect the majority of post procedure pneumothoraces for biopsies in the chest. Post procedural CT will be performed according to the physician's consideration. ** Note ** If any complications are observed while using the ActiSight System, the investigator will revert to using standard procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older at the time of enrollment
* Subjects meeting all medical conditions for percutaneous aspiration/biopsy with safe path to lesion
* INR <1.4
* Written informed consent to participate in the study
* Ability to comply with the requirements of the study procedures

Exclusion Criteria:

* Hemophilia, thrombocytopenia, coagulopathy, or other elevated risk for bleeding or abnormal clotting
* Use of Aspirin or similar antithrombotic medication
* Pulmonary hypertension, heart failure, renal failure, or blood dyscrasia
* Subjects who cannot tolerate mild sedation
* Subjects with the following laboratory values, unless approved by hematologist:

  * Platelet count < 60,000/mL
  * APTT > 39 sec or PT > 15 sec, INR > 1.4
  * Pregnancy or lactation
  * Patient is unable to comply with requirements of the procedure, i.e. holding breath
  * Participation in an investigational trial within 30 days of enrollment
  * Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder, or any chronic condition that could, in the opinion of the investigator, of interfering with the conduct of the study.
  * Subjects who are uncooperative or cannot follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Frequency of target reached (tip of the needle location) within a radius of 8 mm from the preplanned targeted point as measured on the final CT scan | During procedure

SECONDARY OUTCOMES:
Number of needle punctures through the skin | During procedure
Number of CT scans needed | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Liat Appelbaum, Dr., Principal Investigator — Hadassah Ein Carem
Locations (1):
- ActiViews Ltd, Haifa, Israel